CLINICAL TRIAL: NCT02419417
Title: A Phase I/IIa Trial With BMS-986158, a Small Molecule Inhibitor of the Bromodomain and Extra-Terminal (BET) Proteins, as Monotherapy or in Combination With Nivolumab in Subjects With Selected Advanced Solid Tumors or Hematologic Malignancies
Brief Title: Study of BMS-986158 in Subjects With Select Advanced Cancers
Acronym: BET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA011-001; 2015-000324-29 (EudraCT Number)
Record Dates: First submitted 2015-04-02; First posted 2015-04-17 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Advanced Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Treatment (Experimental): Patients treated at various doses and schedules
  Interventions: Drug: BMS-986158
- Combination Therapy (Experimental): Patients treated at selected doses and schdules
  Interventions: Drug: BMS-986158; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986158 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Combination Therapy

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of BMS-986158 in subjects with select advanced cancers

ELIGIBILITY:
Inclusion Criteria:

* Must have select advanced cancers with specific genetic profiles
* Must have received appropriate standard of care
* At least one measurable lesion at baseline
* Expected to have life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) of 0 to 1

Exclusion Criteria:

* Concomitant second malignancies
* Uncontrolled or significant cardiovascular disease
* Inadequate bone marrow function
* Chronic gastrointestinal illness
* Prior treatment with Bromodomain and Extra-Terminal (BET) inhibitor

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (6):
  - City Of Hope National Medical Center, Duarte, California
  - University Of Colorado, Aurora, Colorado
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon
  - Univ. Of Pa, Philadelphia, Pennsylvania
  - Institute for Translational Oncology Research-ITOR, Greenville, South Carolina
- Nucleus Network, Melbourne, Victoria, Australia
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada
- France (2):
  - Local Institution, Lyon
  - Local Institution, Villejuif
- Spain (3):
  - H. Univ. Vall dHebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Clinica Universidad de Navarra, Pamplona

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 participants were treated.
Groups:
- Part 1 Schedule A - BMS-986158 0.75 mg: Single dose of BMS-986158 at 0.75 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
- Part 1 Schedule A - BMS-986158 1.25 mg: Single dose of BMS-986158 at 1.25 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
- Part 1 Schedule A - BMS-986158 2 mg: Single dose of BMS-986158 at 2 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
- Part 1 Schedule A - BMS-986158 3 mg: Single dose of BMS-986158 at 3 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
- Part 1 Schedule A - BMS-986158 4.5 mg: Single dose of BMS-986158 at 4.5 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
- Part 1 Schedule B - BMS-986158 2 mg: Single dose of BMS-986158 at 2 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 14 consecutive days, followed by a 7 days rest period, on a 21 days cycle
- Part 1 Schedule B - BMS-986158 3 mg: Single dose of BMS-986158 at 3 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 14 consecutive days, followed by a 7 days rest period, on a 21 days cycle
- Part 1 Schedule C - BMS-986158 2 mg: Single dose of BMS-986158 at 2 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 7 consecutive days, followed by a 14 days rest period, on a 21 days cycle
- Part 1 Schedule C - BMS-986158 3 mg: Single dose of BMS-986158 at 3 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 7 consecutive days, followed by a 14 days rest period, on a 21 days cycle
- Part 1 Schedule C - BMS-986158 4.5 mg: Single dose of BMS-986158 at 4.5 mg. Approximately 7 days later, BMS-986158 is administered at the same dose QD for 7 consecutive days, followed by a 14 days rest period, on a 21 days cycle
- Part 2 Schedule A: BMS-986158 administered at 4.5 mg QD for 5 consecutive days, followed by a 2 days resting period, for a total of 10 doses.
  Then, BMS-986158 is administered at the 3.75 mg dose QD for 5 consecutive days, followed by a 2 days rest period, on a 28 days cycle
Period: Overall Study
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Started | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Not completed — Disease progression | 5 | 4 | 13 | 10 | 10 | 3 | 4 | 5 | 13 | 9 | 0
Not completed — Study drug toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event unrelated to study drug | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Participant request to discontinue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A | Total
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 7 | 7 | 10 | 3 | 2 | 6 | 12 | 7 | 1 | 63
  >=65 years | 1 | 0 | 6 | 3 | 3 | 1 | 2 | 0 | 1 | 3 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (7.2) | 45.0 (9.4) | 63.2 (12.1) | 54.3 (16.4) | 55.5 (15.4) | 61.3 (3.0) | 68.5 (5.4) | 58.8 (2.7) | 53.6 (9.1) | 58.1 (9.9) | 30.0 (NA) — Only 1 participant was treated in this arm | 57.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 12 | 7 | 9 | 2 | 3 | 5 | 9 | 9 | 0 | 64
  Male | 0 | 1 | 1 | 3 | 4 | 2 | 1 | 1 | 4 | 1 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 0 | 1 | 6 | 6 | 5 | 2 | 2 | 4 | 4 | 6 | 1 | 37
  Unknown or Not Reported | 5 | 3 | 7 | 4 | 8 | 2 | 2 | 1 | 8 | 3 | 0 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 5 | 3 | 11 | 10 | 10 | 4 | 4 | 6 | 8 | 8 | 0 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4 | 1 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing different types of events, including Adverse Events (AEs), Serious Adverse Events (SAEs), AEs leading to discontinuation and deaths.
  Events are classified based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose to 30 days following last dose (up to approximately 29 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Participants
  Adverse Events (AEs) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 9 | 1
  Serious Adverse Events (SAEs) | 3 | 3 | 7 | 7 | 9 | 2 | 2 | 4 | 5 | 3 | 0
  AEs leading to discontinuation | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0
  Deaths | 0 | 1 | 2 | 4 | 3 | 0 | 0 | 1 | 2 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Hepatic Test Values
Description: Number of participants experiencing abnormal hepatic function, as measured by different parameters.
  ALT = Alanine aminotransferase AST = Aspartate aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days following last dose (up to approximately 29 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Participants
  ALT OR AST > 3XULN | 2 | 1 | 2 | 2 | 2 | 0 | 1 | 0 | 2 | 2 | 0
  ALT OR AST > 5XULN | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0
  ALT OR AST > 10XULN | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 1
  CONCURRENT ALT OR AST > 3XULN AND BILIRUB > 2XULN WITHIN 1 DAY | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  CONCURRENT ALT OR AST > 3XULN AND BILIRUB > 2XULN WITHIN 30 DAYS | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR, as assessed by the investigator, is defined as the best response designation, recorded between the dates of first dose and the date of first objectively documented progression (per RECIST v1.1 for solid tumors, Lugano 2014 criteria for hematologic malignancies or PCWG3 for prostate cancer) or the date of subsequent therapy, whichever occurs first.
Time Frame: From first dose to date of first documented progression or subsequent therapy (up to approximately 28 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Stable Disease | 1 | 1 | 2 | 1 | 7 | 2 | 1 | 1 | 4 | 4 | 0
  Progressive Disease | 4 | 2 | 8 | 7 | 3 | 2 | 2 | 2 | 9 | 4 | 0
  Unable to determine | 0 | 1 | 3 | 2 | 2 | 0 | 1 | 3 | 0 | 2 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR)
Time Frame: From first dose to date of first documented progression or subsequent therapy (up to approximately 28 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Percent of Participants | 0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 0 [0.0 to 24.7] | 0 [0.0 to 30.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 45.9] | 0 [0.0 to 24.7] | 0 [0.0 to 30.8] | 100.0 [2.5 to 100.0]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time between the date of first response and the date of the first objectively documented disease progression (as determined by RECIST v1.1 for solid tumors, Lugano 2014 criteria for hematologic malignancies, or PCWG3 (including PSA assessments) for prostate cancer [CRPC or NEPC]), or death due to any cause, whichever occurs first.
Time Frame: From date of first response to date of first objectively documented disease progression or death (up to approximately 42 weeks)
Population: All participants who achieved a Complete Response (CR) or Partial Response (PR)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weeks |  |  |  |  | 22.3 (NA) — Only 1 participant was analyzed in this cohort |  |  |  |  |  | 42.4 (NA) — Only 1 participant was analyzed in this cohort

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the first dose of study medication to the date of the first objective documentation of tumor progression or death due to any cause.
Time Frame: From first dose to date of first objectively documented disease progression or death (up to approximately 28 months)
Population: All treated participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Weeks | 4.57 [2.86 to 14.43] | 9.71 [6.57 to 25.43] | 7.57 [3.57 to 15.86] | 7.43 [2.57 to 8.43] | 13.79 [5.14 to 24.57] | 24.29 [6.29 to 120.14] | 6.57 [5.57 to 40.14] | 8.29 [5.29 to NA] — Insufficient number of events | 8.43 [7.43 to 13.29] | 9.14 [4.57 to 18.14] | NA [NA to NA] — Insufficient number of events

7. Secondary Outcome: Progression Free Survival Rate (PFSR)
Description: PFSR is defined as the percentage of participants who remain progression free and surviving at the specified timepoints (12 weeks, 24 weeks, and 48 weeks).
  Reported values are estimates derived from Kaplan-Meier analyses
Time Frame: From first dose to 12 weeks, to 24 weeks, and to 48 weeks after first dose
Population: All treated participants.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
Number analyzed (Participants) | 5 | 4 | 13 | 10 | 13 | 4 | 4 | 6 | 13 | 10 | 1
Percent of participants
  12 weeks | 20.0 [0.8 to 58.2] | 33.3 [0.9 to 77.4] | 27.3 [6.5 to 53.9] | 11.1 [0.6 to 38.8] | 50.0 [18.4 to 75.3] | 50.0 [5.8 to 84.5] | 33.3 [0.9 to 77.4] | 20.0 [0.8 to 58.2] | 27.5 [6.6 to 54.2] | 45.7 [11.0 to 75.7] | 100.0 [100.0 to 100.0]
  24 weeks | 0.0 [NA to NA] — Insufficient number of events | 33.3 [0.9 to 77.4] | 9.1 [0.5 to 33.3] | 11.1 [0.6 to 38.8] | 30.0 [7.1 to 57.8] | 50.0 [5.8 to 84.5] | 33.3 [0.9 to 77.4] | 0.0 [NA to NA] — Insufficient number of events | 18.3 [2.9 to 44.4] | 0.0 [NA to NA] — Insufficient number of events | 100.0 [100.0 to 100.0]
  48 weeks | 0.0 [NA to NA] — Insufficient number of events | 0.0 [NA to NA] — Insufficient number of events | 0.0 [NA to NA] — Insufficient number of events | 0.0 [NA to NA] — Insufficient number of events | 0.0 [NA to NA] — Insufficient number of events | 25.0 [0.9 to 66.5] | 0.0 [NA to NA] — Insufficient number of events | 0.0 [NA to NA] — Insufficient number of events | 9.2 [0.5 to 33.5] | 0.0 [NA to NA] — Insufficient number of events | 100.0 [100.0 to 100.0]

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Single Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- BMS-986158 0.75 mg: All participants treated with BMS-986158 at 0.75 mg dose, regardless of the dosing schedule.
- BMS-986158 1.25 mg: All participants treated with BMS-986158 at 1.25 mg dose, regardless of the dosing schedule.
- BMS-986158 2 mg: All participants treated with BMS-986158 at 2 mg dose, regardless of the dosing schedule.
- BMS-986158 3 mg: All participants treated with BMS-986158 at 3 mg dose, regardless of the dosing schedule.
- BMS-986158 4.5 mg: All participants treated with BMS-986158 at 4.5 mg dose, regardless of the dosing schedule.
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 16 | 25 | 17
ng/mL
  Parent BMS-986158 | 68.8 (23) | 175 (36) | 269 (25) | 368 (30) | 513 (25)
  Metabolite BMT-161485: number analyzed (Participants) | 5 | 3 | 15 | 24 | 17
  Metabolite BMT-161485 | 5.00 (30) | 10.0 (29) | 18.2 (36) | 21.6 (47) | 35.6 (41)

9. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) - Single Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 16 | 25 | 17
Hours
  Parent BMS-986158 | 4.00 [2.00 to 4.02] | 1.00 [1.00 to 2.00] | 1.04 [0.500 to 4.03] | 1.02 [0.500 to 6.15] | 2.02 [1.00 to 4.03]
  Metabolite BMT-161485: number analyzed (Participants) | 5 | 3 | 15 | 24 | 17
  Metabolite BMT-161485 | 24.0 [2.55 to 24.2] | 2.00 [2.00 to 24.0] | 6.00 [1.00 to 72.0] | 3.03 [0.983 to 48.0] | 6.27 [1.00 to 48.0]

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve in One Dosing Interval (AUC(0-24)) - Single Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 16 | 25 | 17
hr*ng/mL
  Parent BMS-986158 | 1027 (16) | 2309 (13) | 3533 (25) | 4989 (38) | 7039 (34)
  Metabolite BMT-161485: number analyzed (Participants) | 5 | 3 | 15 | 24 | 17
  Metabolite BMT-161485 | 98.2 (34) | 188 (11) | 310 (35) | 377 (44) | 629 (41)

11. Secondary Outcome: Apparent Terminal Phase Half-Life (T-HALF) - Single Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 3 | 11 | 18 | 14
hr
  Parent BMS-986158 | 33.7 (1.41) | 48.7 (6.66) | 54.3 (19.87) | 42.7 (19.56) | 43.8 (15.75)
  Metabolite BMT-161485: number analyzed (Participants) | 1 | 3 | 8 | 11 | 10
  Metabolite BMT-161485 | 35.3 (NA) — Only 1 participants analyzed in this cohort | 50.8 (6.26) | 48.8 (18.78) | 39.4 (13.80) | 38.7 (13.66)

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) - Single Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 3 | 11 | 18 | 14
hr*ng/mL
  Parent BMS-986158 | 2479 (18) | 7013 (17) | 9775 (56) | 11677 (44) | 18974 (40)
  Metabolite BMT-161485: number analyzed (Participants) | 1 | 3 | 8 | 11 | 10
  Metabolite BMT-161485 | 409 (NA) — Only 1 participants analyzed in this cohort | 892 (13) | 944 (73) | 1128 (46) | 2231 (67)

13. Secondary Outcome: Apparent Total Body Clearance (CLT/F) - Single Dose Administration
Description: Values are reported only for the parent BMS-986158
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 16 | 25 | 17
mL/min | 5.04 (17) | 2.97 (18) | 3.41 (56) | 4.28 (62) | 3.95 (33)

14. Secondary Outcome: Apparent Volume of Distribution of Terminal Phase (Vz/F) - Single Dose Administration
Description: Values are reported only for the parent BMS-986158
Time Frame: From drug administration in Cycle 1 Day 1 to 168 hours post drug administration
Population: All treated participants with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | BMS-986158 0.75 mg | BMS-986158 1.25 mg | BMS-986158 2 mg | BMS-986158 3 mg | BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 3 | 11 | 18 | 14
Liters | 14.7 (21) | 12.5 (18) | 14.8 (27) | 14.4 (28) | 14.1 (31)

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Multiple Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485.
  Values are also reported separately for Cycle 1 Day 1 and the latest collection timepoint available (Cycle 2 Day 5 for Schedule A, Cycle 2 day 14 for Schedule B, Cycle 2 Day 7 for Schedule C)
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: All treated participants with available measurements. PK data not collected for the participant in Part 2 Schedule A cohort
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
ng/mL
  Parent BMS-986158 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
  Parent BMS-986158 - Cycle 1 Day 1 | 68.8 (23) | 175 (36) | 260 (20) | 328 (36) | 478 (24) | 207 (NA) — Only 1 participant analyzed in this cohort | 481 (25) | 295 (29) | 370 (22) | 567 (24)
  Parent BMS-986158 - Latest timepoint: number analyzed (Participants) | 4 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - Latest timepoint | 136 (43) | 284 (16) | 442 (29) | 624 (44) | 898 (39) | 279 (NA) — Only 1 participant analyzed in this cohort | 855 (NA) — Only 1 participant analyzed in this cohort | 520 (34) | 588 (47) | 901 (62)
  Metabolite BMT-161485 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Metabolite BMT-161485 - Cycle 1 Day 1 | 5.00 (30) | 10.0 (29) | 16.9 (32) | 22.5 (38) | 30.0 (41) | 13.6 (NA) — Only 1 participant analyzed in this cohort | 26.3 (63) | 21.1 (35) | 19.4 (44) | 45.5 (32)
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 25.8 (82) | 31.0 (25) | 49.4 (46) | 83.3 (57) | 126 (50) | 32.7 (NA) — Only 1 participant analyzed in this cohort | 127 (NA) — Only 1 participant analyzed in this cohort | 80.7 (53) | 64.5 (55) | 146 (83)

16. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) - Multiple Dose Administration
Description: as for outcome 15
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
Hours
  Parent BMS-986158 - Cycle 1 day 1: number analyzed (Participants) | 5 | 3 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
  Parent BMS-986158 - Cycle 1 day 1 | 4.00 [2.00 to 4.02] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.03] | 2.00 [0.983 to 6.15] | 2.04 [1.00 to 4.03] | 1.00 [1.00 to 1.00] | 1.03 [1.00 to 4.03] | 1.00 [0.500 to 2.03] | 1.00 [0.500 to 2.02] | 2.02 [1.00 to 4.00]
  Parent BMS-986158 - Latest timepoint: number analyzed (Participants) | 4 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - Latest timepoint | 3.14 [2.00 to 6.05] | 1.50 [0.500 to 2.00] | 2.00 [0.500 to 4.02] | 2.01 [0.500 to 2.10] | 2.00 [1.00 to 4.05] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [0.833 to 4.00] | 1.66 [0.967 to 2.03] | 2.00 [0.167 to 2.03]
  Metabolite BMT-161485 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Metabolite BMT-161485 - Cycle 1 Day 1 | 24.0 [2.55 to 24.2] | 2.00 [2.00 to 24.0] | 5.08 [2.00 to 72.0] | 23.9 [0.983 to 48.0] | 15.1 [1.00 to 48.0] | 1.00 [1.00 to 1.00] | 1.52 [1.00 to 47.4] | 14.9 [1.00 to 71.5] | 2.02 [1.00 to 48.0] | 6.27 [1.00 to 45.6]
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 24.0 [24.0 to 24.0] | 4.00 [1.50 to 6.00] | 2.07 [0 to 4.02] | 2.01 [1.00 to 6.10] | 4.00 [1.00 to 24.0] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 4.08 [3.83 to 24.0] | 4.00 [0 to 6.32] | 4.00 [1.00 to 27.1]

17. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) - Multiple Dose Administration
Description: as for outcome 15
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
h*ng/mL
  Parent BMS-986158 - Cycle 1 day 1: number analyzed (Participants) | 5 | 3 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
  Parent BMS-986158 - Cycle 1 day 1 | 2150 (15) | 6372 (14) | 8564 (48) | 10452 (50) | 19124 (46) | 5202 (NA) — Only 1 participant analyzed in this cohort | 25852 (41) | 10931 (43) | 11493 (54) | 17220 (84)
  Parent BMS-986158 - Latest timepoint: number analyzed (Participants) | 4 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - Latest timepoint | 3449 (93) | 4961 (73) | 7612 (71) | 13378 (77) | 29517 (36) | 6321 (NA) — Only 1 participant analyzed in this cohort | 33978 (NA) — Only 1 participant analyzed in this cohort | 19868 (45) | 18266 (97) | 19995 (135)
  Metabolite BMT-161485 - Cycle 1 day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Metabolite BMT-161485 - Cycle 1 day 1 | 314 (32) | 790 (14) | 992 (65) | 1305 (48) | 2748 (64) | 424 (NA) — Only 1 participant analyzed in this cohort | 2467 (61) | 1895 (58) | 1219 (73) | 2645 (77)
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 1474 (89) | 691 (73) | 1110 (89) | 2925 (85) | 6691 (49) | 1000 (NA) — Only 1 participant analyzed in this cohort | 7339 (NA) — Only 1 participant analyzed in this cohort | 5022 (62) | 3458 (96) | 5719 (134)

18. Secondary Outcome: Area Under the Plasma Concentration-Time Curve in One Dosing Interval (AUC(0-24)) - Multiple Dose Administration
Description: as for outcome 15
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
h*ng/mL
  Parent BMS-986158 - Cycle 1 day 1 | 1027 (16) | 2309 (13) | 3610 (22) | 4942 (43) | 6786 (24) | 2358 (NA) — Only 1 participant analyzed in this cohort | 6921 (28) | 3660 (27) | 4468 (29) | 7418 (43)
  Parent BMS-986158 - Latest timepoint: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - Latest timepoint | 2716 (51) | 3852 (NA) — Only 1 participant analyzed in this cohort |  | 9817 (56) | 14551 (32) | 3430 (NA) — Only 1 participant analyzed in this cohort | 13305 (NA) — Only 1 participant analyzed in this cohort | 8561 (36) | 8637 (71) | 11286 (104)
  Metabolite BMT-161485 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Metabolite BMT-161485 - Cycle 1 Day 1 | 98.2 (34) | 188 (11) | 290 (22) | 404 (39) | 560 (42) | 191 (NA) — Only 1 participant analyzed in this cohort | 439 (52) | 367 (36) | 337 (46) | 741 (38)
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 550 (81) | 500 (NA) — Only 1 participant analyzed in this cohort |  | 1746 (64) | 2649 (48) | 505 (NA) — Only 1 participant analyzed in this cohort | 2551 (NA) — Only 1 participant analyzed in this cohort | 1765 (51) | 1299 (63) | 2616 (102)

19. Secondary Outcome: Minimum Observed Concentration Within a Dosing Interval (Cmin) - Multiple Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485.
  Values are reported only for the latest collection timepoint available (Cycle 2 Day 5 for Schedule A, Cycle 2 day 14 for Schedule B, Cycle 2 Day 7 for Schedule C)
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
ng/mL
  Parent BMS-986158 - Latest timepoint | 73.7 (45) | 141 (17) | 208 (53) | 227 (76) | 428 (41) | 85.1 (NA) — Only 1 participant analyzed in this cohort | 435 (NA) — Only 1 participant analyzed in this cohort | 270 (42) | 238 (94) | 253 (125)
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 16.4 (91) | 22.3 (22) | 33.7 (55) | 54.0 (73) | 89.6 (55) | 14.4 (NA) — Only 1 participant analyzed in this cohort | 79.5 (NA) — Only 1 participant analyzed in this cohort | 59.7 (54) | 44.2 (74) | 71.1 (115)

20. Secondary Outcome: Concentration at the End of Dosing Interval (C24) - Multiple Dose Administration
Description: as for outcome 15
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
ng/mL
  Parent BMS-986158 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 9 | 10 | 10 | 1 | 4 | 6 | 11 | 7
  Parent BMS-986158 - Cycle 1 Day 1 | 33.5 (18) | 67.4 (12) | 108 (36) | 143 (50) | 210 (32) | 66.1 (NA) — Only 1 participant analyzed in this cohort | 232 (30) | 112 (33) | 125 (43) | 185 (68)
  Parent BMS-986158 - Latest timepoint: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - Latest timepoint | 87.9 (63) | 116 (NA) — Only 1 participant analyzed in this cohort |  | 280 (64) | 461 (36) | 85.1 (NA) — Only 1 participant analyzed in this cohort | 463 (NA) — Only 1 participant analyzed in this cohort | 276 (45) | 244 (93) | 263 (131)
  Metabolite BMT-161485 - Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Metabolite BMT-161485 - Cycle 1 Day 1 | 4.85 (29) | 7.92 (8) | 12.0 (37) | 18.8 (40) | 27.0 (44) | 5.23 (NA) — Only 1 participant analyzed in this cohort | 19.0 (42) | 16.3 (37) | 12.9 (58) | 29.1 (53)
  Metabolite BMT-161485 -Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 -Latest timepoint | 16.4 (91) | 22.3 (22) | 33.7 (55) | 54.0 (73) | 89.6 (55) | 14.4 (NA) — Only 1 participant analyzed in this cohort | 104 (NA) — Only 1 participant analyzed in this cohort | 69.4 (62) | 47.8 (74) | 84.5 (120)

21. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough) - Multiple Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485.
  Values are also reported separately for the first and last collection
Time Frame: From Cycle (C)2 Day (D)2 to C2D5 (Schedule A) or from C2D14 to C4D8 (Schedule B) or from C2D7 to C8D8 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 3 | 4 | 8 | 9 | 1 | 1 | 3 | 6 | 7
ng/mL
  Parent BMS-986158 - First collection | 35.7 (25) | 79.6 (10) | 142 (51) | 138 (48) | 257 (27) | 109 (NA) — Only 1 participant analyzed in this cohort | 435 (NA) — Only 1 participant analyzed in this cohort | 242 (58) | 282 (98) | 284 (119)
  Parent BMS-986158 -Last collection: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 0 | 1 | 1 | 0
  Parent BMS-986158 -Last collection | 87.9 (63) | 116 (NA) — Only 1 participant analyzed in this cohort |  | 280 (64) | 461 (36) | 289 (NA) — Only 1 participant analyzed in this cohort |  | 69.1 (NA) — Only 1 participant analyzed in this cohort | 370 (NA) — Only 1 participant analyzed in this cohort |
  Metabolite BMT-161485 - First collection | 7.78 (36) | 9.42 (19) | 11.4 (51) | 22.2 (48) | 36.5 (44) | 16.9 (NA) — Only 1 participant analyzed in this cohort | 79.5 (NA) — Only 1 participant analyzed in this cohort | 51.2 (68) | 49.4 (81) | 75.3 (110)
  Metabolite BMT-161485 - Last collection: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 0 | 1 | 1 | 0
  Metabolite BMT-161485 - Last collection | 25.8 (82) | 20.1 (NA) — Only 1 participant analyzed in this cohort |  | 65.8 (63) | 108 (47) | 36.4 (NA) — Only 1 participant analyzed in this cohort |  | 10.8 (NA) — Only 1 participant analyzed in this cohort | 24.5 (NA) — Only 1 participant analyzed in this cohort |

22. Secondary Outcome: Accumulation Index (AI) - Multiple Dose Administration
Description: AI is defined as the ratio of an exposure measure at steady-state to that after the first dose. Reported exposure measures include Cmax, C24 and AUC24.
  Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485.
Time Frame: Cycle 2 Day 5 (Schedule A) or Cycle 2 Day 14 (Schedule B) or Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 3 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
Ratio
  Parent BMS-986158 - Cmax | 1.89 (20) | 1.72 (20) | 1.76 (34) | 1.94 (42) | 1.79 (29) | 1.35 (NA) — Only 1 participant analyzed in this cohort | 2.37 (NA) — Only 1 participant analyzed in this cohort | 1.65 (13) | 1.50 (38) | 1.59 (47)
  Parent BMS-986158 - C24: number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - C24 | 2.58 (51) |  |  | 1.79 (38) | 2.24 (29) | 1.29 (NA) — Only 1 participant analyzed in this cohort | 3.05 (NA) — Only 1 participant analyzed in this cohort | 2.55 (24) | 1.98 (54) | 1.42 (72)
  Parent BMS-986158 - AUC24: number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Parent BMS-986158 - AUC24 | 2.60 (35) |  |  | 1.95 (38) | 2.15 (23) | 1.45 (NA) — Only 1 participant analyzed in this cohort | 2.78 (NA) — Only 1 participant analyzed in this cohort | 2.34 (22) | 1.90 (46) | 1.52 (59)
  Metabolite BMT-161485 - Cmax: number analyzed (Participants) | 3 | 3 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 - Cmax | 4.53 (54) | 3.44 (38) | 2.91 (27) | 3.46 (33) | 4.45 (30) | 2.40 (NA) — Only 1 participant analyzed in this cohort | 6.35 (NA) — Only 1 participant analyzed in this cohort | 4.12 (36) | 3.08 (59) | 3.21 (64)
  Metabolite BMT-161485 - C24: number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 - C24 | 4.63 (58) |  |  | 3.18 (38) | 4.33 (39) | 2.76 (NA) — Only 1 participant analyzed in this cohort | 6.23 (NA) — Only 1 participant analyzed in this cohort | 4.46 (31) | 4.02 (42) | 2.91 (79)
  Metabolite BMT-161485 - AUC24: number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Metabolite BMT-161485 - AUC24 | 5.06 (45) |  |  | 4.20 (55) | 5.03 (34) | 2.64 (NA) — Only 1 participant analyzed in this cohort | 6.85 (NA) — Only 1 participant analyzed in this cohort | 4.66 (25) | 3.87 (54) | 3.53 (87)

23. Secondary Outcome: Effective Elimination Half-Life (Effective T-HALF) - Multiple Dose Administration
Description: Values are reported separately for the parent BMS-986158 and its metabolite BMT-161485.
Time Frame: Cycle 2 Day 5 (Schedule A) or Cycle 2 Day 14 (Schedule B) or Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
Hours
  Parent BMS-986158: number analyzed (Participants) | 3 | 0 | 0 | 7 | 8 | 1 | 1 | 5 | 7 | 5
  Parent BMS-986158 | 36.0 (15.99) |  |  | 25.7 (14.86) | 27.3 (8.72) | 14.4 (NA) — Only 1 participant analyzed in this cohort | 37.3 (NA) — Only 1 participant analyzed in this cohort | 31.6 (10.48) | 27.3 (15.15) | 27.6 (19.11)
  Metabolite BMT-161485 | 80.9 (40.42) |  |  | 72.1 (47.11) | 80.4 (29.59) | 35.2 (NA) — Only 1 participant analyzed in this cohort | 105 (NA) — Only 1 participant analyzed in this cohort | 72.7 (19.42) | 63.5 (39.53) | 72.8 (74.17)

24. Secondary Outcome: Ratio of Metabolite (BMT-161485) Maximum Observed Plasma Concentration (Cmax) to Parent (BMS-986158) Cmax - Multiple Dose Administration
Description: Values are reported separately for Cycle 1 Day 1 and the latest collection timepoint available (Cycle 2 Day 5 for Schedule A, Cycle 2 day 14 for Schedule B, Cycle 2 Day 7 for Schedule C)
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
Ratio
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Cycle 1 Day 1 | 0.073 (0.0104) | 0.057 (0.0052) | 0.068 (0.0204) | 0.078 (0.0268) | 0.068 (0.0303) | 0.066 (NA) — Only 1 participant analyzed in this cohort | 0.059 (0.0247) | 0.077 (0.0373) | 0.056 (0.0187) | 0.083 (0.0209)
  Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Latest timepoint | 0.179 (0.0726) | 0.112 (0.0329) | 0.115 (0.0290) | 0.144 (0.0528) | 0.142 (0.0260) | 0.117 (NA) — Only 1 participant analyzed in this cohort | 0.149 (NA) — Only 1 participant analyzed in this cohort | 0.163 (0.0536) | 0.115 (0.0371) | 0.173 (0.0576)

25. Secondary Outcome: Ratio of Metabolite (BMT-161485) Area Under the Plasma Concentration-Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) to Parent (BMS-986158) AUC(0-T) - Multiple Dose Administration
Description: as for outcome 24
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 4 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
Ratio
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
  Cycle 1 Day 1 | 0.154 (0.0504) | 0.127 (0.0369) | 0.125 (0.0262) | 0.152 (0.0572) | 0.151 (0.0558) | 0.081 (NA) — Only 1 participant analyzed in this cohort | 0.099 (0.0279) | 0.182 (0.0632) | 0.114 (0.0473) | 0.170 (0.0821)
  Latest timepoint: number analyzed (Participants) | 3 | 4 | 7 | 8 | 8 | 1 | 1 | 5 | 8 | 7
  Latest timepoint | 0.247 (0.1000) | 0.141 (0.0248) | 0.150 (0.0377) | 0.234 (0.0787) | 0.233 (0.0558) | 0.158 (NA) — Only 1 participant analyzed in this cohort | 0.216 (NA) — Only 1 participant analyzed in this cohort | 0.274 (0.1184) | 0.203 (0.0788) | 0.320 (0.1552)

26. Secondary Outcome: Ratio of Metabolite (BMT-161485) Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) to Parent (BMS-986158) AUC(INF) - Multiple Dose Administration
Time Frame: Cycle 1 Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 1 | 3 | 4 | 4 | 5 | 1 | 1 | 3 | 6 | 5
Ratio | 0.177 (NA) — Only 1 participant analyzed in this cohort | 0.131 (0.0426) | 0.120 (0.0286) | 0.158 (0.0307) | 0.164 (0.0809) | 0.080 (NA) — Only 1 participant analyzed in this cohort | 0.106 (NA) — Only 1 participant analyzed in this cohort | 0.139 (0.0401) | 0.103 (0.0357) | 0.184 (0.0947)

27. Secondary Outcome: Ratio of Metabolite (BMT-161485) Area Under the Plasma Concentration-Time Curve in One Dosing Interval (AUC(0-24)) to Parent (BMS-986158) AUC(0-24) - Multiple Dose Administration
Description: as for outcome 24
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 5 (Schedule A) or to Cycle 2 Day 14 (Schedule B) or to Cycle 2 Day 7 (Schedule C)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 5 | 3 | 8 | 9 | 10 | 1 | 4 | 6 | 11 | 7
Ratio
  Cycle 1 Day 1 | 0.099 (0.0290) | 0.081 (0.0055) | 0.086 (0.0208) | 0.097 (0.0425) | 0.087 (0.0347) | 0.081 (NA) — Only 1 participant analyzed in this cohort | 0.066 (0.0221) | 0.102 (0.0178) | 0.080 (0.0283) | 0.108 (0.0445)
  Latest timepoint: number analyzed (Participants) | 3 | 1 | 0 | 7 | 8 | 1 | 1 | 5 | 8 | 7
  Latest timepoint | 0.213 (0.0786) | 0.130 (NA) — Only 1 participant analyzed in this cohort |  | 0.192 (0.0697) | 0.187 (0.0475) | 0.147 (NA) — Only 1 participant analyzed in this cohort | 0.192 (NA) — Only 1 participant analyzed in this cohort | 0.218 (0.0770) | 0.160 (0.0561) | 0.253 (0.1151)

28. Secondary Outcome: Change From Baseline in Electrocardiogram Parameter QTcF
Description: QT Interval corrected for Fridericia's Formula. Change from baseline is calculated from pre-dose at the indicated timepoints.
Time Frame: From Cycle 1 Day 1 to last dosing day in Cycle 2 (C2D8 for Schedule A, C2D14 for Schedule B, C2D7 for Schedule C).
Population: All treated participants with available measurements at the indicated timepoints. PK data not collected for the participant in Part 2 Schedule A cohort
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg
Number analyzed (Participants) | 4 | 1 | 9 | 8 | 11 | 3 | 1 | 4 | 8 | 8
msec | -6.8 (11.63) | -5.3 (NA) — Only 1 participant analyzed in this cohort | -3.3 (22.48) | -5.4 (18.45) | -10.2 (22.43) | -10.7 (15.10) | -16.7 (NA) — Only 1 participant analyzed in this cohort | -7.7 (10.98) | 14.3 (14.03) | -0.6 (10.75)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 68 months). Serious Adverse events and other adverse events were assessed from date of first dose to 30 days following date of last dose (up to approximately 29 months).
Description: All treated participants
Arm/Group | Part 1 Schedule A - BMS-986158 0.75 mg | Part 1 Schedule A - BMS-986158 1.25 mg | Part 1 Schedule A - BMS-986158 2 mg | Part 1 Schedule A - BMS-986158 3 mg | Part 1 Schedule A - BMS-986158 4.5 mg | Part 1 Schedule B - BMS-986158 2 mg | Part 1 Schedule B - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 2 mg | Part 1 Schedule C - BMS-986158 3 mg | Part 1 Schedule C - BMS-986158 4.5 mg | Part 2 Schedule A
All-Cause Mortality (participants affected / at risk) | 5/5 | 3/4 | 10/13 | 8/10 | 12/13 | 3/4 | 3/4 | 4/6 | 10/13 | 7/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/4 | 7/13 | 7/10 | 9/13 | 2/4 | 2/4 | 4/6 | 5/13 | 3/10 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 12/13 | 10/10 | 13/13 | 4/4 | 4/4 | 6/6 | 13/13 | 9/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Schedule A - BMS-986158 0.75 mg (N=5) | Part 1 Schedule A - BMS-986158 1.25 mg (N=4) | Part 1 Schedule A - BMS-986158 2 mg (N=13) | Part 1 Schedule A - BMS-986158 3 mg (N=10) | Part 1 Schedule A - BMS-986158 4.5 mg (N=13) | Part 1 Schedule B - BMS-986158 2 mg (N=4) | Part 1 Schedule B - BMS-986158 3 mg (N=4) | Part 1 Schedule C - BMS-986158 2 mg (N=6) | Part 1 Schedule C - BMS-986158 3 mg (N=13) | Part 1 Schedule C - BMS-986158 4.5 mg (N=10) | Part 2 Schedule A (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Schedule A - BMS-986158 0.75 mg (N=5) | Part 1 Schedule A - BMS-986158 1.25 mg (N=4) | Part 1 Schedule A - BMS-986158 2 mg (N=13) | Part 1 Schedule A - BMS-986158 3 mg (N=10) | Part 1 Schedule A - BMS-986158 4.5 mg (N=13) | Part 1 Schedule B - BMS-986158 2 mg (N=4) | Part 1 Schedule B - BMS-986158 3 mg (N=4) | Part 1 Schedule C - BMS-986158 2 mg (N=6) | Part 1 Schedule C - BMS-986158 3 mg (N=13) | Part 1 Schedule C - BMS-986158 4.5 mg (N=10) | Part 2 Schedule A (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 9 | 1 | 2 | 1 | 4 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 6 | 8 | 2 | 4 | 0 | 5 | 3 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 5 | 0 | 4 | 1 | 0 | 2 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6 | 7 | 10 | 3 | 2 | 4 | 8 | 7 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 8 | 3 | 7 | 1 | 0 | 6 | 7 | 5 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 7 | 2 | 6 | 1 | 1 | 5 | 5 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 2 | 3 | 0 | 2 | 1 | 3 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 4 | 10 | 3 | 5 | 4 | 1 | 2 | 5 | 5 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 4 | 0 | 2 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Suprapubic pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 2 | 2 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation retinopathy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 1 | 5 | 2 | 0 | 1 | 3 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 6 | 3 | 7 | 2 | 2 | 3 | 3 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 5 | 2 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 2 | 4 | 2 | 0 | 2 | 3 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 5 | 2 | 1 | 0 | 6 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02419417/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02419417/SAP_001.pdf